CLINICAL TRIAL: NCT02877043
Title: Measurement of the Quality: Application to Lung Resection for Cancer Using a National PMSI Database
Brief Title: Study of the Quality of Lung Resection
Acronym: ResPul
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PAGES AOI 2015
Record Dates: First submitted 2016-08-04; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Bronchial Cancer
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients undergoing lung resection
  Interventions: Procedure: resection pulmonaire

INTERVENTIONS:
Procedure: resection pulmonaire

SUMMARY:
In 2009, centres that carried out lung resection for cancer were required to obtain authorization following the first cancer plan. One of the criteria to obtain authorization was the volume of activity: the centre had to carry out at least 30 lung resections per year for cancer. Five years later, it would be useful to know the impact of this new organization of oncology on the quality of care. To answer this question, the PMSI database is an ideal source of an indicator of quality: in-hospital mortality. This observational cohort study will be conducted using the national PMSI database with data covering the period from 1st January 2005 to 31st December 2013. It will be limited to hospitalization for lung resection. The time will be divided into 3 periods: 2005-2007, 2008-2010 and 2011-2013; the period 2008-2010 includes the implementation of authorizations for cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

Any patients who underwent lung resection for bronchial cancer will be included in this study. The PMSI (Programme de Médicalisation des Systèmes d'Information) database will be searched for all patients with:

* A principal diagnosis of ICD10 (international classification of diseases) codes for bronchial cancer
* And CCAM (Classification Commune des Actes médicaux ) procedure codes for lung resection (segmentectomy, lobectomy, pneumonectomy).

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing lung resection
Sampling Method: Non-Probability Sample
Enrollment: 72000 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
number of deaths during hospitalization | 9 years
  number of death during hospitalization for pulmonary resection from 2005 to 2013

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France